CLINICAL TRIAL: NCT00240097
Title: Study of Sequential Topoisomerase, Irinotecan/Oxaliplatin-Etoposide/Carboplatin in Extensive SCLC
Brief Title: Study of Sequential Topoisomerase, Irinotecan/Oxaliplatin - Etoposide /Carboplatin in Extensive Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Sanofi-Synthelabo (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor of Medicine, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F041222002; UAB 0421 (Other: institutional protocol study number)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Oxaliplatin; pegfilgrastim; Irinotecan; Carboplatin; Etoposide; etoposide phosphate; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irinotecan; Oxaliplatin; Neulasta (Experimental): Irinotecan (I.V.) 150-200 mg/m2; Day 1 (every 5 weeks) Oxaliplatin (I.V.) 85 mg/m2; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 1 (every 5 weeks)
  Interventions: Drug: Intervention A: Irinotecan; Oxaliplatin; Neulasta
- Etoposide; Carboplatin; Neulasta (Experimental): Etoposide (I.V.) 100 mg/m2; Day 1, 2, 3 (every 5 weeks) Carboplatin (I.V.) area under the concentration curve (AUC) 6; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 4 (every 5 weeks)
  Interventions: Drug: Intervention B: Etoposide; Carboplatin; Neulasta

INTERVENTIONS:
Drug: Intervention A: Irinotecan; Oxaliplatin; Neulasta — Irinotecan (I.V.) 150-200 mg/m2; Day 1 (every 5 weeks) Oxaliplatin (I.V.) 85 mg/m2; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 1 (every 5 weeks)
  Other Names: Camptosar; Eloxatin; Pegfilgrastim
  Arms: Irinotecan; Oxaliplatin; Neulasta
Drug: Intervention B: Etoposide; Carboplatin; Neulasta — Etoposide (I.V.) 100 mg/m2; Day 1, 2, 3 (every 5 weeks) Carboplatin (I.V.) AUC 6; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 4 (every 5 weeks)
  Other Names: VP-16; Etopophos®; Vepesid®; Taxol; Paraplatin; Pegfilgrastim
  Arms: Etoposide; Carboplatin; Neulasta

SUMMARY:
The primary objective of Part I of the study is to determine tumor response rate of sequential topoisomerase targeting with irinotecan/oxaliplatin followed by etoposide /carboplatin in chemotherapy-naïve patients with extensive small cell lung cancer. The primary objective of Part II of the study is to determine the objective tumor response rate of irinotecan/oxaliplatin in patients with either refractory disease or who have relapsed to first line chemotherapy or chemoradiotherapy.

DETAILED DESCRIPTION:
This is a Phase II, open label study for either chemotherapy-naïve patients with extensive SCLC or patients who are refractory or have relapsed to 1st line therapy for SCLC. The primary objective is to determine the objective response rate.

This study consists of 2 parts:

Part I - Chemotherapy-naïve patients with extensive SCLC

• These patients will be treated with sequential topoisomerase targeting regimens (Regimen A and B). Regimen A consists of irinotecan and oxaliplatin (IROX), given on Day 1, and Neulasta administered on Day 2. Regimen B consists of etoposide and carboplatin, given on Day 15(etoposide will be given daily x 3)and Neulasta on Day 18. Then, Regimen A will be given again 3 weeks later. The first re-evaluation for response will be performed 3 weeks after the second round of the sequential regimens.

Schema of Part I:

Regimen A (→ 2 weeks) Regimen B (→ 3 weeks) Regimen A (→ 2 weeks) Regimen B → (3 weeks) → Re-Stage

* The second re-evaluation for response will be performed 3 weeks after the fourth round of the sequential regimen. At this point patients with stable disease will be observed; those with either a partial or complete response will be treated with another round of sequential therapy (Regimen A → Regimen B) if there is no evidence of unacceptable toxicity. At the end (3 weeks after) of the fifth round of chemotherapy, patients will be re-evaluated for response, and will be followed-up for recurrent disease every 8 weeks.
* Analysis of Top I and Top II levels in peripheral blood mononuclear cells will be performed in 10 patients of Part I.
* Evaluation of the expression of the ERCC genes (ERCC1, ERCC2, and XPF) will be performed in those patients in Part I with an adequate tumor specimen.

Part II - Patients who have either refractory disease or have relapsed from 1st line therapy

• These patients will be treated with Regimen A1 (IROX) at 3-week intervals. Neulasta will be administered on Day 2 of each cycle. The first re-evaluation for response will be performed 3 weeks after the 3rd cycle of Regimen A1. The second re-evaluation for response will be performed 3 weeks after the 6th cycle of Regimen A1. At this point, patients with stable disease will be observed; those with either a partial or complete response will be treated with two additional cycles of Regimen A1 if there is no evidence of unacceptable toxicity. At the end (3 weeks after) of the 8th cycle of Regimen A1, patients will be re-evaluated for response, and will be followed-up for recurrent disease every 8 weeks.

Schema of Part II:

Regimen A1 (→ 3 weeks) Regimen A1 (→ 3 weeks) Regimen A1 (→ 3 weeks) Re-Stage

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of SCLC.
2. Measurable or assessable tumor parameters.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
4. Age between 18 and 79 years (in the State of Alabama > 18).
5. Adequate bone marrow, liver and renal function, defined as:

   * Absolute neutrophil count (ANC) ≥ 1500/µL
   * Platelet count ≥ 100,000/µL
   * SGOT/SGPT ≤ 2.5 x upper limit of normal or ≤ 5 x upper limit of normal when liver metastases are present.
   * Total bilirubin value ≤ 1.5 x upper limit of normal.
   * Serum creatinine value ≤ 1.5 x upper limit of normal.
6. Fully recovered from any previous surgery (at least 4 weeks since major surgery)
7. Must have recovered from prior radiation therapy (at least 3 weeks)
8. All participants must agree to practice approved methods of birth control (if applicable). A negative pregnancy test must be documented during the screening period for women of childbearing potential.
9. Must provide written informed consent and authorization to use and disclose health information (HIPAA).

   For Part I
10. Extensive-stage SCLC as defined as disease not confined to one hemithorax, including ipsilateral pleural effusion or pericardial effusion.
11. No prior chemotherapy.

    For Part II
12. Patients with either refractory disease, or who have relapsed 1st line therapy. No prior chemotherapy with Oxaliplatin or irinotecan.
13. Demonstrated tumor progression at the time of study entry.

Exclusion Criteria:

1. Concurrent cancer chemotherapy, biologic therapy or radiotherapy.
2. Administration of any investigational drug within 28 days prior to administration of the current therapy.
3. Symptomatic brain metastases; those patients should be treated first with either whole brain radiation therapy or radiosurgery.
4. Concurrent serious infection.
5. Concomitant severe or uncontrolled underlying medical disease unrelated to the tumor, which is likely to compromise patient safety and affect the outcome of the study.
6. History of other malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for a minimum of 2 years.
7. Neuropathy at baseline ≥ Grade 2.
8. Any evidence or history of hypersensitivity or other contraindications for the drugs used in this trial.
9. History of chronic diarrhea; or diarrhea (excess of 2-3 stools/day above normal frequency) in the past 2 weeks.
10. History of a positive serology for human immunodeficiency virus (HIV).
11. Psychiatric disorder that prevents patients from providing informed consent or following protocol instructions.
12. Pregnant or lactating women.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Rossman J, Reddy V, Cantor A, Miley D, Robert F. Phase II study of dose-intense chemotherapy with sequential topoisomerase-targeting regimens with irinotecan/oxaliplatin followed by etoposide/carboplatin in chemotherapy naive patients with extensive small cell lung cancer. Lung Cancer. 2011 May;72(2):219-23. doi: 10.1016/j.lungcan.2010.08.023. Epub 2010 Oct 8. PMID 20934233

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A and B: Regimen A Irinotecan (I.V.) 150-200 mg/m2; Day 1 (every 5 weeks) Oxaliplatin (I.V.) 85 mg/m2; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 1 (every 5 weeks)
  Regimen B Etoposide (I.V.) 100 mg/m2; Day 1, 2, 3 (every 5 weeks) Carboplatin (I.V.) AUC 6; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 4 (every 5 weeks)
Period: Part I
Arm/Group | Regimen A and B
Started | 30
Completed | 26
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — histology | 1
Not completed — unevaluable | 1
Period: Part II
Arm/Group | Regimen A and B
Started | 26
Completed | 3
Not Completed | 23
Not completed — did not continue from Part I | 23

BASELINE CHARACTERISTICS:
Groups:
- Regimen A and B: Chemotherapy-naive patients with extensive SCLC will be treated in one of two regimens: Regimen A consists of treatment with irinotecan and oxaliplatin given every 2 weeks while Regimen B consists of etoposide and carboplatin given every 3 weeks. Both regimens will include re-evaluation for response at least every 8 weeks.
Arm/Group | Regimen A and B
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Secondary Outcome: Progression Free Survival (Part I)
Description: Time to progressive disease
Time Frame: baseline to five years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regimen A and B
Number analyzed (Participants) | 26
months | 8.95 [6.5 to 9.8]

2. Primary Outcome: Objective Response Rate (Part I)
Description: The primary objective is to determine the objective tumor response rate of sequential topoisomerase targeting with irinotecan/oxaliplatin followed by etoposide/carboplatin in chemotherapy-naïve patients with extensive SCLC and Stage IIIb (wet) - IV Large Cell Carcinoma of the Lung with neuroendocrine markers. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Stable response means did not meet criteria for progressive or partical response. 20% progressive disease.
Time Frame: baseline to 18 months
Measure: Number; unit: Participants
Arm/Group | Regimen A and B
Number analyzed (Participants) | 26
Participants
  Complete response | 4
  Partial response | 20
  Stable disease | 1
  Progressive disease | 0
  Unevaluable | 1

3. Secondary Outcome: Overall Survival (Part I)
Description: Length of subject survival after starting study treatment
Time Frame: baseline to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regimen A and B
Number analyzed (Participants) | 26
months | 12.9 [10.2 to 15.5]

4. Primary Outcome: Response Rate After Relapse
Description: The objective is to determine the objective tumor response rate of sequential topoisomerase targeting with irinotecan/oxaliplatin followed by etoposide/carboplatin in chemotherapy-naïve patients with extensive SCLC and Stage IIIb (wet) - IV Large Cell Carcinoma of the Lung with neuroendocrine markers. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Stable response means did not meet criteria for progressive or partical response. 20% progressive disease.
Time Frame: 3 weeks after 3rd cycle of starting therapy after relapse or refractory disease
Population: All subjects dropped out or died prior to experiencing relapse
Groups:
- Part II - After Relapse: Study dosing with A and B based on relapse
Arm/Group | Part II - After Relapse
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Regimen A First Cycle; Regimen A Overall Toxicity: Regimen A Irinotecan (I.V.) 150-200 mg/m2; Day 1 (every 5 weeks) Oxaliplatin (I.V.) 85 mg/m2; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 1 (every 5 weeks)
- Regimen B First Cycle; Regimen B Overall Toxicity: Regimen B Etoposide (I.V.) 100 mg/m2; Day 1, 2, 3 (every 5 weeks) Carboplatin (I.V.) AUC 6; Day 1 (every 5 weeks) Neulasta (subcutaneous) 6 mg; Day 4 (every 5 weeks)
Arm/Group | Regimen A First Cycle | Regimen B First Cycle | Regimen A Overall Toxicity | Regimen B Overall Toxicity
Serious Adverse Events (participants affected / at risk) | 3/26 | 6/26 | 7/26 | 19/26
Other Adverse Events (participants affected / at risk) | 7/26 | 6/26 | 20/26 | 13/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A First Cycle (N=26) | Regimen B First Cycle (N=26) | Regimen A Overall Toxicity (N=26) | Regimen B Overall Toxicity (N=26)
Grade 3 Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 19 (24)
Grade 4 Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0) | 15 (22)
Grade 3 Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (9)
Grade 3 nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Grade 3 diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (6) | 0 (0)
Grade 3 Fatigue (General disorders) | 1 (1) | 1 (1) | 5 (6) | 2 (2)
Grade 3 Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (4) | 1 (1)
Grade 4 Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (6) | 2 (3) | 6 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A First Cycle (N=26) | Regimen B First Cycle (N=26) | Regimen A Overall Toxicity (N=26) | Regimen B Overall Toxicity (N=26)
nausea and vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 12 (16) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 7 (9) | 1 (1)
Fatigue (General disorders) | 7 (7) | 6 (6) | 20 (29) | 13 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No